CLINICAL TRIAL: NCT05667584
Title: Comparisons of the Blood Pressure Control Ability Between Hypotension Prediction Index With Non-invasive Continuous Arterial Pressure Waveforms, Continuous Blood Pressure Monitoring With Non-invasive Continuous Arterial Pressure Waveforms, and Intermittent Blood Pressure Monitoring With Conventional Non-invasive Blood Pressureduring Neuraxial Anesthesia in Cesarean Section: a Randomized Controlled Trial
Brief Title: Comparisons of Blood Pressure Control Ability Between HPI, ClearSight, and Conventional NIBP During Neuraxial Anesthesia in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202210114RINC
Record Dates: First submitted 2022-12-11; First posted 2022-12-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2022-12

CONDITIONS: Intraoperative Hypotension; Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HPI (Experimental): Standard intraoperative monitor and non-invasive continuous arterial pressure waveforms (ClearSight) are set up in this group. ClearSight data and hypotension prediction index (HPI) derived from ClearSight are used for recording and monitoring. Blood pressure is monitored with ClearSight and HPI. Attending anesthesiologists controlled the blood pressure according to HPI values.
  1. Maintain HPI below 85
  2. HPI > 85 and heart rate > 60/min, IV bolus norepinephrine 5-10 mcg
  3. HPI > 85 and heart rate < 60/min, IV bolus norepinephrine 5-10 mcg with atropine 0.01 mg/kg
  Interventions: Device: hypotension prediction index derived from non-invasive arterial pressure waveforms
- ClearSight (Active Comparator): Standard intraoperative monitor and non-invasive continuous arterial pressure waveforms (ClearSight) are set up in this group. ClearSight data and HPI derived from ClearSight are used for recording, and HPI are masked for attending anesthesiologists. Blood pressure is monitored with ClearSight. Attending anesthesiologists controlled the blood pressure according to continuous arterial pressure values.
  1. Maintain mean arterial pressure (MAP) above 65 mmHg
  2. MAP < 65mmHg and heart rate > 60/min, IV bolus norepinephrine 5-10 mcg
  3. MAP < 65mmHg and heart rate < 60/min, IV bolus norepinephrine 5-10 mcg with atropine 0.01 mg/kg
  Interventions: Device: non-invasive arterial pressure waveforms
- NIBP (No Intervention): Standard intraoperative monitor and non-invasive continuous arterial pressure waveforms (ClearSight) are set up in this group. ClearSight data and HPI derived from ClearSight are used for recording, and are masked for attending anesthesiologists. Blood pressure is monitored with conventional non-invasive blood pressure (NIBP). Attending anesthesiologists controlled the blood pressure according to continuous arterial pressure values.
  1. Maintain mean arterial pressure (MAP) above 65 mmHg
  2. MAP < 65mmHg and heart rate > 60/min, IV bolus norepinephrine 5-10 mcg
  3. MAP < 65mmHg and heart rate < 60/min, IV bolus norepinephrine 5-10 mcg with atropine 0.01 mg/kg

INTERVENTIONS:
Device: hypotension prediction index derived from non-invasive arterial pressure waveforms — The Hypotension Prediction Index (HPI) is an algorithm based on the complex analysis of features in high-fidelity arterial pressure waveform recordings developed to observe subtle signs that could predict the onset of hypotension in surgical and intensive care unit patients. HPI is a unitless number that ranges from 1 to 100, and as the number increases, the likelihood of a hypotensive event (MAP <65 mm Hg for more than 1 minute) occurring in the near future increases. In a validation study on HPI conducted in patients under general anesthesia, the algorithm, at its optimal value, predicted hypotension with both sensitivity and specificity of 86% 5 minutes before the event. Measurement of the arterial pressure waveforms using a finger cuff (ClearSight) is well established.
  Arms: HPI
Device: non-invasive arterial pressure waveforms — ClearSight is a non-invasive hemodynamic monitoring device using digital-cuff and volume-clamp technology to obtain a continuous arterial blood pressure waveform. Continuous finger blood pressure measurement is established by wrapping the cuff around the middle phalanx of a finger. The area under the waveform curve is analyzed using a unique algorithm that serves to calculate the arterial blood pressure, stroke volume (SV) and CO.
  Arms: ClearSight

SUMMARY:
The goal of this study is to compare the blood pressure control ability with HPI, ClearSight, and conventional NIBP during neuraxial anesthesia in cesarean section. The main question it aims to answer is:

Anesthesiologists can have a better control of blood pressure during cesarean section with HPI than with conventional NIBP.

During the surgery, the participants will be monitored with standard monitor and HPI with ClearSight and will be randomly assigned to three groups, including HPI group, ClearSight group, and NIBP group. Anesthesiologists will treat intraoperative hypotension with different protocols according to the participants' allocation. Investigators will compare the time-weighted average mean arterial pressure < 65mmHg with in three groups. Secondary outcomes includes the intraoperative hypotension rate, total duration of hypotension, the hypotension symptoms and signs of parturients.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 50 year-old parturients
* scheduled cesarean delivery
* neuraxial anesthesia

Exclusion Criteria:

* parturients with preeclampsia
* parturients with cardiovascular disease above NYHA functional class 2
* parturients with arrhythmias, preoperative severe hypertension, or other severe cardiopulmonary diseases.
* severe perioperative arrhythmias with or without hemodynamic instability
* failed neuraxial anesthesia or regional blockade level below T6

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
time-weighted MAP below 65 mmHg | through the surgery completion, an average of 1.5 hours

SECONDARY OUTCOMES:
rates of parturients with intraoperative hypotension | through the surgery completion, an average of 1.5 hours
  hypotension is defined as MAP below 65 mmHg for more than 1 minute
total hypotension duration | through the surgery completion, an average of 1.5 hours
  hypotension is defined as MAP below 65 mmHg for more than 1 minute
area under curve of hypotension | through the surgery completion, an average of 1.5 hours
  hypotension is defined as MAP below 65 mmHg for more than 1 minute
total vasopressor dosage | through the surgery completion, an average of 1.5 hours
  average norepinephrine dosage used during the surgery
rate of hypotension related symptoms and sign of the parturients | through the surgery completion, an average of 1.5 hours
  symptoms and signs include nausea, vomiting, bradycardia, dizziness, and shivering
average regional cerebral oxygen saturation | through the surgery completion, an average of 1.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Frassanito L, Sonnino C, Piersanti A, Zanfini BA, Catarci S, Giuri PP, Scorzoni M, Gonnella GL, Antonelli M, Draisci G. Performance of the Hypotension Prediction Index With Noninvasive Arterial Pressure Waveforms in Awake Cesarean Delivery Patients Under Spinal Anesthesia. Anesth Analg. 2022 Mar 1;134(3):633-643. doi: 10.1213/ANE.0000000000005754. PMID 34591796
- [Background] Misugi T, Juri T, Suehiro K, Kitada K, Kurihara Y, Tahara M, Hamuro A, Nakano A, Koyama M, Mori T, Tachibana D. Non-invasive continuous blood pressure monitoring using the ClearSight system for pregnant women at high risks of post-partum hemorrhage: comparison with invasive blood pressure monitoring during cesarean section. Obstet Gynecol Sci. 2022 Jul;65(4):325-334. doi: 10.5468/ogs.22063. Epub 2022 Jun 27. PMID 35754365